CLINICAL TRIAL: NCT05679336
Title: Rituximab, Cyclophosphamide, and Corticosteroids at Low Cumulative Doses to Induce Remission in Primary Membranous Nephropathy
Brief Title: Rituximab, Cyclophosphamide, and Corticosteroids in Primary Membranous Nephropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VD-266/MN
Record Dates: First submitted 2022-11-28; First posted 2023-01-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Membranous Nephropathy - PLA2R Induced
Keywords: Rituximab; Corticosteroids; Cyclophosphamide; Clinical and immunological remissions; Membranous nephropathy; Nephrotic syndrome
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrotic Syndrome | interventions — Rituximab; Cyclophosphamide; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab, Cyclophosphamide, and Corticosteroids group (Experimental): The experimental treatment group: 40 participants will receive combined immunosuppressive therapy with Rituximab, Cyclophosphamide, and Corticosteroids.
  Interventions: Drug: Rituximab, Cyclophosphamide, and Corticosteroids

INTERVENTIONS:
Drug: Rituximab, Cyclophosphamide, and Corticosteroids — 1. Rituximab (RTX) will be given as a single intravenous (IV) dose of 375 mg/m2. Extra RTX infusion at the same dose will be administered on weeks 12, 24, and 36 in the absence of remission and the occurrence of peripheral B-cell reconstitution. Peripheral B-cell reconstitution is defined as total CD19+ cell count >5 cells/μL;
  2. Concurrent with RTX initiation, a single IV infusion of methylprednisolone 500 mg will be administrated, followed by oral prednisolone 1 mg/kg daily but not exceeding 60 mg daily during week 1. The dosage will be rapidly decreased by 10 mg/weekly as follows: week 2, 50 mg daily; week 3, 40 mg daily; week 4, 30 mg daily; week 5, 20 mg daily; weeks 6-7, 10 mg daily; weeks 8-48, 5 mg daily; week 49, stop;
  3. Four IV infusions of Cyclophosphamide will be administered at a dose of 7.5 mg/kg every other week (on weeks 1, 3, 5, and 7).

SUMMARY:
This exploratory study aims to assess the efficacy, safety of the experimental treatment based on a combination of rituximab (RTX), intravenous (IV) cyclophosphamide (CYC), and corticosteroids (S) administrated at lower cumulative doses (RCP) for the induction of early remission in subjects with anti-PLA2R antibody-positive primary membranous nephropathy (PMN) having nephrotic syndrome (NS).

DETAILED DESCRIPTION:
BACKGROUND

PMN is a glomerular disease associated with autoantibodies targeting podocyte antigens, mostly the phospholipase A2 receptor (anti-PLA2R). The formation of subepithelial immune complexes and complement-mediated injury to podocyte and glomerular basement membrane leads, in most cases, to the development of NS and the risk of its life-threatening complications: thromboembolic, infectious, and metabolic. Standard renoprotective approaches are not sufficient for many patients with PMN and persistent NS. In randomized clinical trials of immunosuppressive therapies, up to 68% of patients failed to achieve remission during the first 12 months without substantial differences in efficacy between immunosuppressive regimens. Treatment failures are increased in high-risk patients, including those with heavier proteinuria and higher serum anti-PLA2R levels. As a result, a significant proportion of patients remain for a long time at high risk of severe complications due to persistent high-level proteinuria and NS, and disease progression.

PROPOSED NEW TREATMENT APPROACH

Collectively, in the past decades no significant progress has been achieved in the treatment of patients with PMN, and up to 40% of the patients still progress to dialysis. In this context, therapies that may result in a higher response and lower relapse rates at an acceptable rate of adverse effects are warranted. Particularly, developing of treatment approaches to rapid induction of remission is critically important to prevent life-threatening NS complications, stop disease progression, and improve long-term prognosis, especially in high-risk patients.

We conducted a pilot open-label trial in 14 patients (mean age 51±12 years, men - 70%) with PMN and NS and high serum level of anti-PLA2R treated with RTX, CYC and S. The overall remission was achieved in 100% of cases (of which complete remissions (CR) in 21.4%) with the median time-to-remission of 2.5 (1.0; 3.5) months. The most commonly observed side effects were infusion related (flu-like symptoms, chills/rigors, fever, fatigue, headache, hypotension,) and typically responded to antihistamines. No patient, except one, had a major drug-related adverse event in 15.7 patient-years. This adverse event was transient elevation of transaminases in induction phase, leading to several days delay in administration of next dose of CYC and prolongation of hospital stay. Thus, according to these results, the use of multi-targeted therapy with RTX, CYC, and S at low dosages seems to be an effective approach for the rapid induction of PMN remission and prevention of NS complications.

The study population will comprise of adult male and female subjects aged 18 - 75 years with a biopsy-proven PMN, positive for serum anti-PLA2R antibodies. Biopsy-proven PMN defined upon the exclusion of any significant concomitant disease (infectious, autoimmune, neoplastic) by careful clinical work-up at the time of kidney biopsy. Most of patients are expected to have high or very high risk of disease progression according to current KDIGO guidelines.

STUDY DESIGN

This exploratory single-center study aims to assess the efficacy, safety of treatment based on a combination of RTX, IV CYC, and S administrated at lower cumulative doses (RCP) for the induction of early remission in subjects with anti-PLA2R antibody-positive PMN having NS and high risk of progression. Subjects meeting the inclusion criteria and agreed to experimental treatment will be treated with the RCP regimen, and will be prospectively followed. During the study, we plan to do an interim analysis to confirm an expected efficacy and safety of the experimental treatment. Besides analyzing the experimental treatment group itself regarding primary and secondary end-points, we plan to compare to the RCP group two age- and gender-matched historic control groups. Control group 1 will include patients treated with Cyclosporine (CSA) in combination with S, and control group 2 will include patients with treatment based on RTX infusions either as monotherapy or in combination with CSA. Both controls will have to fulfill same eligibility criteria. These comparisons will allow to assess whether the RCP protocol may have an advantage over standard treatments based on RTX or CSA in primary and secondary efficacy criteria: early remission rate, the time to clinical and immunological remissions, and the change in proteinuria, serum albumin and estimated GFR by CKD-EPI equation (eGFR).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Biopsy-proven primary membranous nephropathy (PMN) defined upon the exclusion of any significant concomitant disease (infectious, autoimmune, neoplastic) by careful clinical work-up at the time of kidney biopsy.
3. Signed informed consent
4. Increased serum level of anti-PLA2R antibodies (>20 RU/ml).
5. Absence of contraindications to immusuppressive therapy.
6. Presence of nephrotic syndrome (NS) with one of the following conditions:

   1. persistence for >6 months despite treatment with an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker with or without immunosuppression and NS complications.
   2. persistence for <6 months at the presence of complications related to NS (thromboembolic or infectious event or estimated GFR by CKD-EPI equation (eGFR) decrease >20%.
   3. recurrence after remission with a prior immunosuppressive treatment.
   4. treatment failure of an alternative immunosuppressive regimen.

Exclusion Criteria:

1. Presence of a secondary cause of membranous nephropathy (e.g. hepatitis B, systemic lupus erythematosus, medications, malignancies).
2. Presence of Type 1 or 2 diabetes mellitus: to exclude proteinuria secondary to diabetic nephropathy.
3. Acute or chronic infection, including: current use of suppressive therapy for chronic infection, hospitalization for treatment of infection in the past 60 days, or parenteral anti-microbial (including anti-bacterial, anti-viral, or anti- fungal agents) use in the past 60 days for infection.
4. Women of child-bearing potential who are pregnant, nursing, or unwilling to be sexually inactive or use FDA-approved contraception until study week.
5. A history of mental illness (including any history of suicidal behavior in the last 6 months, any suicidal ideation in the last 2 months, or who, in the investigator's judgment, pose a significant suicide risk).
6. A history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or organ transplantation.
7. Vaccination with a live vaccine within the past 30 days.
8. Evidence of current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence in the past 12 months.
9. Inability to comply with study and follow-up procedures.
10. Laboratory tests meeting any of the following: Hemoglobin <80 g/L; Platelet <80 x 109/ L; Neutrophil <1.0×109/ L; Aspartate aminotransferase (AST) or amino acid aminotransferase (ALT) >2.5× upper limit of normal.
11. Any patient judged by the investigator to be ineligible for enrollment in the trial.
12. eGFR ≤30 ml/min/1.73m2 in one measurement performed at baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Partial clinical remission (PR) and complete clinical remission (CR) | Up to 1 year
  Including the proportion of participants with complete and partial responses by month 12 since the treatment initiation; CR defined as proteinuria of <0.3 g/1.73 m2/24h and serum albumin >30 g/l; PR defined as a ≥50% reduction in proteinuria from baseline accompanied by a regress of nephrotic syndrome (NS)
Time to clinical remission | Up to 1 year
  Cumulative rate of overall (complete and partial) clinical remission and complete clinical remission by month 12

SECONDARY OUTCOMES:
The time to immunologic remission | Through study completion, an average of 2 years
  Cumulative proportion of patients with the immunologic remission by month 12 and thereafter
The change in circulating CD19+ cells | Up to 1 year
  Change of circulating CD19+ cells number from baseline by flow cytometry
The change in proteinuria | Up to 1 year
  Change in 24-h proteinuria from baseline
The change in estimated GFR (eGFR) | Through study completion, an average of 2 years
  Change of eGFR by CKD-EPI equation from baseline
The change in serum albumin | Up to 1 year
  Median monthly change of serum albumin from baseline
Disease relapse since the RCP treatment initiation (in experimental group received Rituximab, Cyclophosphamide, and Corticosteroids at low cumulative doses) | Through study completion, an average of 2 years
  Number of patients experienced disease relapse since the RCP treatment initiation; relapse is defined as 24-h proteinuria >3.5 g after achieving CR or, in those with PR, as an increase of proteinuria >50% compared with the lowest value during remission with recurrence of NS.
Adverse events (AEs) | Through study completion, an average of 2 years
  AEs associated with the RCP therapy: serious adverse events (SAEs) will be defined as the US Food and Drug Administration recommended; AEs will be graded based on the NCI Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dobronravov, Professor, Principal Investigator — St. Petersburg State Pavlov Medical University
Locations (1):
- St. Petersburg State Pavlov Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No